CLINICAL TRIAL: NCT00426062
Title: Free Radical Level in SCC of Tongue Patients Tumor, Serum and Saliva
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Other Study IDs: SHEBA-06-4116-AD-CTIL
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Last update posted 2007-02-21 (Estimated); Status verified 2007-02

CONDITIONS: Squamous Cell Carcinoma
Keywords: Squamous Cell Carcinoma of Tongue and mouth floor
MeSH Terms: conditions — Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Study comparing level of free radicals in tumor tissue, blood serum and saliva in patients with Squamous Cell Carcinoma of tongue and mouth floor. Patients with benign fibroma of oral cavity and normal gingiva around extracted lower wisdom tooth are used for control

ELIGIBILITY:
Inclusion Criteria:

1. Older than 18 years of age.
2. Mentally healthy
3. SCC of Tongue or Mouth Floor
4. Benign Fibroma of Oral Cavity
5. Lower wisdom tooth extraction -

Exclusion Criteria:

1. Younger than 18 years of age
2. Mentally incapacitated

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Alex Dobriyan, DMD, Principal Investigator — Sheba Medical Center; Ran Yahalom, DMD, Principal Investigator — Sheba Medical Center; Rafi Nagler, DMD,MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel